CLINICAL TRIAL: NCT06737276
Title: Dietary Advice Training in Nursing Using Simulation and Interactive Fiction: a Randomised Controlled Trial
Brief Title: Dietary Advice Training in Nursing Using Simulation and Interactive Fiction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cadiz (Other)
Responsible Party: Principal Investigator, Antonio Jesús Marín Paz, Principal Investigator, University of Cadiz
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: sol-202200229602-tra
Record Dates: First submitted 2024-12-05; First posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Simulation Training; Computer Simulation; Diet, Food, and Nutrition; Nutrition Assessment; Nutrition Therapy; Education, Nursing; Teaching Innovation
Keywords: Simulation Training; Computer Simulation; Diet, Food, and Nutrition; Nutrition Assessment; Nutrition Therapy; Education, Nursing; Teaching Innovation

STUDY DESIGN:
Intervention Model Description: This study is a two-stage simultaneous parallel (CG) and crossover (EG1 and EG2) randomised controlled trial.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The researchers were blinded concerning the randomisation sequence and the allocation of participants to the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental Group 1 (EG1) (Experimental): Participants received a multimodal intervention (intervention order: interactive fiction activities and role-play simulation).
  Interventions: Other: Interactive fiction activities; Other: Role-play simulation
- Experimental Group 2 (EG2) (Experimental): Participants received a multimodal intervention (intervention order: role-play simulation and interactive fiction activities).
  Interventions: Other: Interactive fiction activities; Other: Role-play simulation
- Control Group (CG) (No Intervention): Participants received a conventional practical teaching based on lectures.

INTERVENTIONS:
Other: Interactive fiction activities — The case studies were prepared using interactive fiction through Twine. Each case simulated a nursing consultation with a patient requiring dietary advice, and the patient's evolution depended on the students' choices. All cases created had similar structures, durations, and difficulties to avoid complexity-related bias. For each circumstance, three possible dietary advice options were offered to the patient: one option that would be ideal, one suitable option, and one unsuitable option.
  Arms: Experimental Group 1 (EG1); Experimental Group 2 (EG2)
Other: Role-play simulation — Role-play activity of the nursing consultation on dietary advice according to Nemec et al. (2021) recommendations. Ten case studies of a nursing consultation on dietary advice involving a nurse and a patient were designed with the consensus of a group of nursing professionals with expertise in food and nutrition, health literacy, and communication. Each student was assigned a role and provided with the necessary information to play their character or understand their patient's context. The information provided was different according to the role assigned. They had to perform a simulation of eight minutes, similar to the time available in the student's primary care consultations in the referral health system. Thus, the patient and the family member had to explain the situation or health problem, the professional would analyse it, and together, they would try to reach a therapeutic agreement. After the consultation, a debriefing was carried out.
  Arms: Experimental Group 1 (EG1); Experimental Group 2 (EG2)

SUMMARY:
The goal of this randomised controlled trial is to evaluate the effectiveness of training nursing students using interactive fiction and role-play simulations as teaching methodologies in improving learning and decision-making competencies related to dietary advice.

ELIGIBILITY:
Inclusion Criteria:

* First year of the Degree in Nursing at a Spanish university who were enrolled in the subject "Food, Nutrition and Dietetics".

Exclusion Criteria:

* Lack of attendance since the beginning of the course.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Learning | Pre-test (0 day), Post-test 1 (30th day), and Post-test 2 (60th day)
  The assessment of the learning level during the intervention was measured by correcting the three unpublished case studies created using the interactive fiction methodology. Each case study consisted of 6 questions with 3 possible answers (1 point for the ideal answer, 0.5 points for the adequate answer and 0 points for the inadequate answer). For readability, the final scores were reconverted proportionally out of 10 before statistical analysis.
Decision-making | Pre-test (0 day), Post-test 1 (30th day), and Post-test 2 (60th day)
  Measurement instrument: Clinical Decision-Making in Nursing Scale (CDMNS). It comprises the search for options or alternatives, information seeking and unbiased assimilation of new information, evaluation and re-evaluation of consequences, and probing of goals and values.
Quality of simulations | Post-test 1 (30th day), and Post-test 2 (60th day)
  Measurement instrument: Simulation Design Scale (SDS). This scale measures students' perceptions of 5 dimensions related to simulation design: information, support, problem-solving, guided feedback and fidelity.

SECONDARY OUTCOMES:
Enjoyable experience | Pre-test (0 day), Post-test 1 (30th day), and Post-test 2 (60th day)
  Measurement instrument: Gameful Experience Gamification (GAMEX) scale. It measures 6 dimensions of students' experience in gamified experiences or environments involving interactive enjoyment mechanisms.
Satisfaction | Post-test 1 (30th day), and Post-test 2 (60th day)
  Measurement instrument: Student Satisfaction and Self-Confidence in Learning Scale (SCLS). It has 5 items on student satisfaction with instructional methods, learning materials and instructors, as well as 8 items on self-confidence in learning.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio-Jesús Marín-Paz, PhD, Principal Investigator — University of Cadiz
Locations (1):
- Faculty of Nursing, Algeciras, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: Yes
All data generated and teaching materials created for the interventions.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Unending.
Access Criteria: All data from this study will be available upon request to the author by correspondence, under justified reasons. The teaching material created for the interventions will be deposited in the university's institutional repository.

REFERENCES:
- [Background] Schulz KF, Altman DG, Moher D; CONSORT Group. CONSORT 2010 statement: updated guidelines for reporting parallel group randomised trials. PLoS Med. 2010 Mar 24;7(3):e1000251. doi: 10.1371/journal.pmed.1000251. PMID 20352064
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Marquez-Hernandez VV, Garrido-Molina JM, Gutierrez-Puertas L, Garcia-Viola A, Aguilera-Manrique G, Granados-Gamez G. How to measure gamification experiences in nursing? Adaptation and validation of the Gameful Experience Scale [GAMEX]. Nurse Educ Today. 2019 Oct;81:34-38. doi: 10.1016/j.nedt.2019.07.005. Epub 2019 Jul 12. PMID 31319349
- [Background] Farres-Tarafa M, Bande D, Roldan-Merino J, Hurtado-Pardos B, Biurrun-Garrido A, Molina-Raya L, Raurell-Torreda M, Casas I, Lorenzo-Seva U. Reliability and validity study of the Spanish adaptation of the "Student Satisfaction and Self-Confidence in Learning Scale" (SCLS). PLoS One. 2021 Jul 23;16(7):e0255188. doi: 10.1371/journal.pone.0255188. eCollection 2021. PMID 34297773
- [Background] Ludin SM. Does good critical thinking equal effective decision-making among critical care nurses? A cross-sectional survey. Intensive Crit Care Nurs. 2018 Feb;44:1-10. doi: 10.1016/j.iccn.2017.06.002. Epub 2017 Jun 26. PMID 28663105
- [Background] Correa-Rodriguez M, Pocovi G, Schmidt-RioValle J, Gonzalez-Jimenez E, Rueda-Medina B. Assessment of dietary intake in Spanish university students of health sciences. Endocrinol Diabetes Nutr (Engl Ed). 2018 May;65(5):265-273. doi: 10.1016/j.endinu.2018.01.005. Epub 2018 Mar 26. English, Spanish. PMID 29599102
- [Background] Nemec R, Brower E, Allert J. A Guide to Implementing Role-Play in the Nursing Classroom. Nurs Educ Perspect. 2021 Nov-Dec 01;42(6):E163-E164. doi: 10.1097/01.NEP.0000000000000678. PMID 32472870
- [Background] Jeffries PR, Rodgers B, Adamson K. NLN Jeffries Simulation Theory: Brief Narrative Description. Nurs Educ Perspect. 2015 Sep-Oct;36(5):292-3. doi: 10.5480/1536-5026-36.5.292. No abstract available. PMID 26521496
- [Background] Dwan K, Li T, Altman DG, Elbourne D. CONSORT 2010 statement: extension to randomised crossover trials. BMJ. 2019 Jul 31;366:l4378. doi: 10.1136/bmj.l4378. PMID 31366597
- [Background] Lo YT, Yang CC, Yeh TF, Tu HY, Chang YC. Effectiveness of immersive virtual reality training in nasogastric tube feeding education: A randomized controlled trial. Nurse Educ Today. 2022 Dec;119:105601. doi: 10.1016/j.nedt.2022.105601. Epub 2022 Oct 12. PMID 36244254
- [Background] Karkada S, Radhakrishnan J, Natarajan J, Matua GA, Kaddoura M. Knowledge and Competency of Novice Nursing Students in Nasogastric Tube Feeding: Is Simulation Better than Case Scenario? Oman Med J. 2019 Nov;34(6):528-533. doi: 10.5001/omj.2019.96. PMID 31745417
- [Background] Bridenbaugh JR, Tomesko J, Sandiford D, Tracey DL. Enteral Nutrition Simulation Workshop Enhances Knowledge and Skills of Graduate Nutrition Students. J Nutr Educ Behav. 2023 Apr;55(4):311-315. doi: 10.1016/j.jneb.2022.11.003. Epub 2023 Jan 18. No abstract available. PMID 36670026
- [Background] Tinoco JDS, Enders BC, Sonenberg A, Lira ALBC. Virtual clinical simulation in nursing education: a concept analysis. Int J Nurs Educ Scholarsh. 2021 Jun 18;18(1). doi: 10.1515/ijnes-2020-0001. PMID 34139113
- [Background] Lei YY, Zhu L, Sa YTR, Cui XS. Effects of high-fidelity simulation teaching on nursing students' knowledge, professional skills and clinical ability: A meta-analysis and systematic review. Nurse Educ Pract. 2022 Mar;60:103306. doi: 10.1016/j.nepr.2022.103306. Epub 2022 Feb 2. PMID 35202957
- [Background] Bordelon CJ, Smith TS, Wood T, Watts P. Simulation to Enhance Communication Skills in Neonatal Nursing Practice. Neonatal Netw. 2020 Nov 1;39(6):347-355. doi: 10.1891/0730-0832/11-T-674. PMID 33318231
- [Background] Lame G, Dixon-Woods M. Using clinical simulation to study how to improve quality and safety in healthcare. BMJ Simul Technol Enhanc Learn. 2020 Mar 4;6(2):87-94. doi: 10.1136/bmjstel-2018-000370. Epub 2018 Sep 29. PMID 32133154
- [Background] Hegland PA, Aarlie H, Stromme H, Jamtvedt G. Simulation-based training for nurses: Systematic review and meta-analysis. Nurse Educ Today. 2017 Jul;54:6-20. doi: 10.1016/j.nedt.2017.04.004. Epub 2017 Apr 19. PMID 28456053
- [Background] Shea A, Brophy L, Nininger J, Abbott M, Wilson L. Nutrition integration across the nursing curriculum: A novel teaching model within a pre-licensure program. J Prof Nurs. 2021 Nov-Dec;37(6):1162-1166. doi: 10.1016/j.profnurs.2021.10.006. Epub 2021 Oct 28. PMID 34887035
- [Background] Gianfrancesco C, Johnson M. Exploring the provision of diabetes nutrition education by practice nurses in primary care settings. J Hum Nutr Diet. 2020 Apr;33(2):263-273. doi: 10.1111/jhn.12720. Epub 2019 Dec 2. PMID 31793070
- [Background] Tangvik RJ, Tell GS, Guttormsen AB, Eisman JA, Henriksen A, Nilsen RM, Ranhoff AH. Nutritional risk profile in a university hospital population. Clin Nutr. 2015 Aug;34(4):705-11. doi: 10.1016/j.clnu.2014.08.001. Epub 2014 Aug 12. PMID 25159298
- [Background] Correia MITD, Perman MI, Waitzberg DL. Hospital malnutrition in Latin America: A systematic review. Clin Nutr. 2017 Aug;36(4):958-967. doi: 10.1016/j.clnu.2016.06.025. Epub 2016 Jul 19. PMID 27499391
- [Background] Xu X, Parker D, Ferguson C, Hickman L. Where is the nurse in nutritional care? Contemp Nurse. 2017 Jun;53(3):267-270. doi: 10.1080/10376178.2017.1370782. No abstract available. PMID 28920553
- [Background] Gan T, Cheng HL, Tse MYM. A systematic review of nurse-led dietary interventions for cancer patients and survivors. Asia Pac J Oncol Nurs. 2021 Dec 29;9(2):81-87. doi: 10.1016/j.apjon.2021.12.013. eCollection 2022 Feb. PMID 35529414
- [Background] Crimarco A, Landry MJ, Gardner CD. Ultra-processed Foods, Weight Gain, and Co-morbidity Risk. Curr Obes Rep. 2022 Sep;11(3):80-92. doi: 10.1007/s13679-021-00460-y. Epub 2021 Oct 22. PMID 34677812
- [Background] Chen Z, Khandpur N, Desjardins C, Wang L, Monteiro CA, Rossato SL, Fung TT, Manson JE, Willett WC, Rimm EB, Hu FB, Sun Q, Drouin-Chartier JP. Ultra-Processed Food Consumption and Risk of Type 2 Diabetes: Three Large Prospective U.S. Cohort Studies. Diabetes Care. 2023 Jul 1;46(7):1335-1344. doi: 10.2337/dc22-1993. PMID 36854188
- [Background] Pagliai G, Dinu M, Madarena MP, Bonaccio M, Iacoviello L, Sofi F. Consumption of ultra-processed foods and health status: a systematic review and meta-analysis. Br J Nutr. 2021 Feb 14;125(3):308-318. doi: 10.1017/S0007114520002688. Epub 2020 Aug 14. PMID 32792031
- [Background] Elizabeth L, Machado P, Zinocker M, Baker P, Lawrence M. Ultra-Processed Foods and Health Outcomes: A Narrative Review. Nutrients. 2020 Jun 30;12(7):1955. doi: 10.3390/nu12071955. PMID 32630022
- [Background] Blanco-Rojo R, Sandoval-Insausti H, Lopez-Garcia E, Graciani A, Ordovas JM, Banegas JR, Rodriguez-Artalejo F, Guallar-Castillon P. Consumption of Ultra-Processed Foods and Mortality: A National Prospective Cohort in Spain. Mayo Clin Proc. 2019 Nov;94(11):2178-2188. doi: 10.1016/j.mayocp.2019.03.035. Epub 2019 Oct 14. PMID 31623843
- [Background] Mazza E, Ferro Y, Pujia R, Mare R, Maurotti S, Montalcini T, Pujia A. Mediterranean Diet In Healthy Aging. J Nutr Health Aging. 2021;25(9):1076-1083. doi: 10.1007/s12603-021-1675-6. PMID 34725664